CLINICAL TRIAL: NCT00757120
Title: SCCOR: Alveolar and Airway Mechanisms for COPD Project 3: Membrane-Type 1 Matrix Metalloproteinase and Extracellular Matrix Metalloproteinase Inducer in Cigarette Smoke-Induced Lung Inflammation and Emphysema Pathogenesis
Brief Title: Biomarkers and Genetic Factors Related to Emphysema
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 577
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Emphysema; Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Cigarette Smoke-Induced Inflammation; EMMPRIN; Matrix Metalloproteinase
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood cells, serum, extracted RNA and DNA, lung fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: This group will include current and former smokers who have emphysema.
- 2: This group will include current and former smokers who do not have emphysema.

SUMMARY:
Emphysema, a common type of chronic obstructive pulmonary disease (COPD), is a long-term lung disease that is usually caused by cigarette smoking. This study will examine both current smokers and former smokers who have emphysema, as well as current and former smokers who do not have emphysema, to determine if certain factors found in the blood are related to the risk of developing emphysema.

DETAILED DESCRIPTION:
COPD is a disease in which the lung is damaged and breathing passages become partly obstructed, making it difficult to breathe. Millions of people in the United States have COPD, and it is the fourth leading cause of death in the country. Symptoms include coughing, excess mucus production, shortness of breath and wheezing. Emphysema and chronic bronchitis are illnesses associated with COPD. Emphysema is usually the result of many years of cigarette smoking, but it remains unknown exactly how cigarette smoking causes emphysema. The purpose of this study is to examine current and former smokers who have emphysema and those who do not have emphysema to determine if certain biomarkers or genetic factors are associated with an increased risk of developing the disease. Specifically, study researchers will examine various genes and two proteins, membrane-type-1 matrix metalloproteinase (MT1-MMP) and extracellular matrix metalloproteinase inducer (EMMPRIN), to determine the role they play in the development of emphysema.

Participants will attend one study visit, which will include a medical history review, a blood collection, lung function testing, a 6-minute walk test, and a chest computed tomography (CT) scan. A portion of blood will be stored for current and future genetic research. Participants will also complete questionnaires to collect information on activities, health, and quality of life. Some participants will be invited to return for a bronchoscopy, which is a procedure that allows a doctor to sample the inside of the lungs. Study researchers will contact all participants at the end of the study to collect follow-up medical information.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Able to read and write English
* At least 30 pack-year smoking history (the equivalent of smoking a pack a day for 30 years)
* Able to participate in the informed consent process
* Relatively stable clinical status for the past six weeks (i.e., no illness in the 6 weeks before study entry)

Inclusion Criteria for Participants with Emphysema:

* Global Initiative for Chronic Obstructive Lung Disease (GOLD) class II, III, or IV COPD, as determined by post-bronchodilator spirometry values OR
* More than minimal emphysema on an acceptable-quality chest CT scan

Inclusion Criteria for Participants without Emphysema:

* GOLD class I COPD or GOLD class 0 (2005 classification), as determined post-bronchodilator spirometry values AND
* No or minimal emphysema on an acceptable-quality chest CT scan

Exclusion Criteria:

* Pregnant
* Prisoner
* Vulnerable populations
* Recent illness (defined as increased cough, sputum production, worsening malaise, or need for unscheduled physician visit in the 6 weeks prior to enrollment)
* Coexisting active chronic inflammatory or collagen vascular disease, immunodeficiency of any kind, non-cutaneous malignancy (melanoma is an exclusion), or previous organ transplant
* Congenital abnormalities of the lung or previous lung surgery
* Known active hepatitis B, hepatitis C, or HIV/AIDS (not prospectively evaluated)
* CT evidence of lung disease other than emphysema (including significant fibrosis, bronchiectasis, consolidation, or indeterminate nodules)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will include current and former smokers who previously participated in the National Lung Screening Trial. Patients will also be recruited from the pulmonary clinic at Washington University School of Medicine Jacqueline Maritz Lung Center, the Barnes Jewish Hospital Pulmonary Rehabilitation Program, the Smoking Cessation Clinic of the Siteman Cancer Center, and the Pulmonary Clinic at St. Louis ConnectCare.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holtzman, MD, Study Director — Pulmonary and Critical Care, Washington University in St. Louis; Steven Brody, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Atkinson JJ, Lutey BA, Suzuki Y, Toennies HM, Kelley DG, Kobayashi DK, Ijem WG, Deslee G, Moore CH, Jacobs ME, Conradi SH, Gierada DS, Pierce RA, Betsuyaku T, Senior RM. The role of matrix metalloproteinase-9 in cigarette smoke-induced emphysema. Am J Respir Crit Care Med. 2011 Apr 1;183(7):876-84. doi: 10.1164/rccm.201005-0718OC. Epub 2010 Nov 5. PMID 21057003